CLINICAL TRIAL: NCT02362646
Title: Safety & Efficacy of Intramyocardial Injection of Mesenchymal Precursor Cells on Myocardial Function in LVAD Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annetine Gelijns (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Annetine Gelijns, Chair, Department of Population Health Science & Policy; Edmond A. Guggenheim Professor of Health Policy; Co-Director, InCHOIR, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 08-1078-0008; 2U01HL088942-07 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Cardiomyopathy; Ventricular Dysfunction
Keywords: Heart Failure; Left Ventricular Assist Device; Heart Transplantation; Cardiomyopathy, Destination Therapy; Cell Therapy; Bridge to Transplant
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Ventricular Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPC Intramyocardial Injection (Experimental): Intramyocardial injections of 150 million MPCs
  Interventions: Biological: MPC Intramyocardial Injection
- Control Solution (Sham Comparator): Intramyocardial injections of 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO
  Interventions: Drug: Control Solution

INTERVENTIONS:
Biological: MPC Intramyocardial Injection — Intramyocardial injection of 150 million mesenchymal precursor cells at the time of LVAD implantation
  Other Names: Mesenchymal Precursor Cell Injection; RevascorTM
  Arms: MPC Intramyocardial Injection
Drug: Control Solution
  Other Names: 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO; Cryoprotective media
  Arms: Control Solution

SUMMARY:
The main purpose of this research is to determine whether injecting mesenchymal precursor cells (MPC) into the heart during surgery to implant a left ventricular assist device (LVAD) is safe. MPCs are normally present in human bone marrow and have been shown to increase the development of blood vessels and new heart muscle cells in the heart. In addition, this research is being done to test whether injecting the MPCs into the heart is effective in improving heart function.

DETAILED DESCRIPTION:
Intramyocardial injection of mesenchymal precursor cells (MPC) in patients with advanced heart failure who are treated with left ventricular assist device (LVAD) implantation may result in a renewable source of proliferating functional cardiomyocytes; induce development of capillaries and larger-size blood vessels to supply oxygen and nutrients to endogenous myocardium and newly-implanted cardiomyocytes; and release factors capable of paracrine signaling.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, inclusive of release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation
* Age 18 years or older
* If the subject or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after procedure
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening
* Admitted to the clinical center at the time of randomization
* Clinical indication and accepted candidate for implantation of an FDA-approved (US sites only) or Health Canada-approved (Canadian sites only) implantable, non-pulsatile LVAD as a bridge to transplantation or for destination therapy.

Exclusion Criteria:

* Planned percutaneous LVAD implantation
* Anticipated requirement for biventricular mechanical support
* Concomitant arrhythmia ablation at time of LVAD implantation

  -- Planned aortic valve intervention for aortic insufficiency at the time of LVAD implantation
* Cardiothoracic surgery within 30 days prior to randomization
* Spontaneous myocardial infarction related to ischemia due to a primary coronary event such as unstable plaque rupture, erosion or dissection within 30 days prior to randomization
* Prior cardiac transplantation, LV reduction surgery, or cardiomyoplasty
* Acute reversible cause of heart failure (e.g. myocarditis, profound hypothyroidism)
* Stroke within 30 days prior to randomization
* Platelet count < 100,000/ul within 24 hours prior to randomization
* Acute infectious process: acute bacterial, fungal, or viral disease OR acute exacerbation of chronic infectious disease such as hepatitis
* Presence of >10% anti-HLA antibody titers with known specificity to MPC donor HLA antigens
* A known hypersensitivity to dimethyl sulfoxide (DMSO), murine, and/or bovine products
* History of a known active malignancy within the past 3 years except for localized prostate cancer, cervical carcinoma in situ, breast cancer in situ, or nonmelanoma skin cancer that has been definitively treated
* Presence of human immunodeficiency virus (HIV)
* Received investigational intervention within 30 days prior to randomization
* Treatment and/or an incomplete follow-up treatment of any investigational cell based therapy within 6 months prior to randomization
* Active participation in other research therapy for cardiovascular repair/regeneration
* Prior recipient of stem precursor cell therapy for cardiac repair
* Pregnant or breastfeeding at time of randomization.
* History of known or suspected hypercoagulable state in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-07; Primary Completion 2018-08-10 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O'Gara, MD, Study Chair — Brigham and Women's Hospital; Richard Weisel, MD, Study Chair — Toronto General Hospital
Locations (19):
- United States (16):
  - University of Southern California, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health Systems, Charlottesville, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie de Quebec (Hopital Laval), Québec, Quebec

REFERENCES:
- [Derived] Yau TM, Pagani FD, Mancini DM, Chang HL, Lala A, Woo YJ, Acker MA, Selzman CH, Soltesz EG, Kern JA, Maltais S, Charbonneau E, Pan S, Marks ME, Moquete EG, O'Sullivan KL, Taddei-Peters WC, McGowan LK, Green C, Rose EA, Jeffries N, Parides MK, Weisel RD, Miller MA, Hung J, O'Gara PT, Moskowitz AJ, Gelijns AC, Bagiella E, Milano CA; Cardiothoracic Surgical Trials Network. Intramyocardial Injection of Mesenchymal Precursor Cells and Successful Temporary Weaning From Left Ventricular Assist Device Support in Patients With Advanced Heart Failure: A Randomized Clinical Trial. JAMA. 2019 Mar 26;321(12):1176-1186. doi: 10.1001/jama.2019.2341. PMID 30912838
- See also: Cardiothoracic Surgical Network Website — http://www.ctsurgerynet.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening started in 2014. First patient randomized in July 2015. Last patient randomized in August 2017.
Groups:
- MPC Intramyocardial Injection: MPC Intramyocardial Injection: Intramyocardial injection of 150 million mesenchymal precursor cells (MPCs) at the time of LVAD implantation
- Control Solution: Control Solution: Intramyocardial injections of 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO
Period: Overall Study
Arm/Group | MPC Intramyocardial Injection | Control Solution
Started | 106 | 53
Completed | 68 | 29
Not Completed | 38 | 24
Not completed — Death | 15 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — received transplant | 21 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MPC Intramyocardial Injection | Control Solution | Total
Number analyzed (Participants) | 106 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.3) | 56.9 (11.7) | 56 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 94 | 47 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 100 | 52 | 152
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 16 | 7 | 23
  White | 82 | 40 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Temporary Weans From LVAD Support Tolerated
Description: functional status, defined by the number of temporary weans from LVAD support tolerated over the 6 months post-randomization. A successful wean is the ability to tolerate temporary weaning from LVAD support for 30 minutes without sustained symptoms of worsening heart failure. Wean failures are defined as inability to tolerate the temporary wean for 30 minutes; death; or patient too unstable, in the judgment of the primary heart failure cardiologist, to tolerate the wean attempt.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: number of weans
Arm/Group | MPC Intramyocardial Injection | Control Solution
Number analyzed (Participants) | 106 | 53
number of weans | 0.61 (0.41) | 0.58 (0.45)

2. Primary Outcome: Number of Participants With Adverse Events
Description: Safety as assessed by number of study intervention-related adverse events
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Control Solution: Intramyocardial injections of 50% Alpha-MEM/42.5% ProFreeze NAO Freezing Medium/7.5% DMSO
  Control Solution
Arm/Group | MPC Intramyocardial Injection | Control Solution
Number analyzed (Participants) | 106 | 53
Participants
  Serious AE | 88 | 44
  Other than Serious AE | 33 | 12

3. Secondary Outcome: Physiologic Assessments
Description: Echocardiographic assessments of the myocardial size and function by transthoracic echocardiography with LVAD at full support, and as tolerated following 6-Minute Walk Test (MWT) while weaned from LVAD support (for patients who tolerate wean from LVAD support for 30 minutes)
Time Frame: up to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Histopathological Assessments of Myocardial Tissue
Time Frame: up to 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Time Frame: up to 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Quality of Life (QoL)
Description: Quality of life will be assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ), a widely used tool in heart failure populations, and the Short Form 12 (SF12), a widely used overall health status measure.
Time Frame: 6 months and 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Hopkins Verbal Learning Test
Description: Cognitive performance will be assessed Hopkins Verbal Learning Test. Neurocognitive testing will be administered by clinical site personnel who have been trained and certified for test administration by the Neurocognitive Core lab personnel.
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Trailmaking Tests A and B
Description: Cognitive performance will be assessed using Trailmaking Tests A and B. Neurocognitive testing will be administered by clinical site personnel who have been trained and certified for test administration by the Neurocognitive Core lab personnel.
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

9. Secondary Outcome: MCG Complex Figures
Description: Cognitive performance will be assessed using the MCG Complex Figures. Neurocognitive testing will be administered by clinical site personnel who have been trained and certified for test administration by the Neurocognitive Core lab personnel.
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Digit Span
Description: as for outcome 9
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Digit Symbol Substitution Test
Description: Cognitive performance will be assessed using the Digit Symbol Substitution Test. Neurocognitive testing will be administered by clinical site personnel who have been trained and certified for test administration by the Neurocognitive Core lab personnel.
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Controlled Oral Word Association
Description: Cognitive performance will be assessed using the Controlled Oral Word Association. Neurocognitive testing will be administered by clinical site personnel who have been trained and certified for test administration by the Neurocognitive Core lab personnel.
Time Frame: 3 months and 12 months
Reporting Status: Not Posted

13. Secondary Outcome: Length of Stay
Description: Length of stay of index hospitalization
Time Frame: up to 12 months
Reporting Status: Not Posted

14. Secondary Outcome: Hospitalizations
Description: Frequency and cause of readmissions
Time Frame: up to 12 months
Reporting Status: Not Posted

15. Secondary Outcome: Hospital Costs
Description: Hospital resource use
Time Frame: up to 12 months
Reporting Status: Not Posted

16. Secondary Outcome: Functional Status
Description: functional status, defined by the number of temporary weans from LVAD support tolerated
Time Frame: up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months for adverse events 12 months for mortality
Description: Trial specific protocol-defined adverse event
Arm/Group | MPC Intramyocardial Injection | Control Solution
All-Cause Mortality (participants affected / at risk) | 15/106 | 8/53
Serious Adverse Events (participants affected / at risk) | 88/106 | 41/53
Other Adverse Events (participants affected / at risk) | 33/106 | 12/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MPC Intramyocardial Injection (N=106) | Control Solution (N=53)
Bleeding (General disorders) | 51 | 28
Sustained ventricular dysrhythmia requiring defibrillation or cardioversion (Cardiac disorders) | 26 | 8
Sustained supraventricular dysrhythmia requiring drug treatment or cardioversion (Cardiac disorders) | 12 | 9
Pump thrombus confirmed (Injury, poisoning and procedural complications) | 10 | 3
Pump thrombus suspected (Injury, poisoning and procedural complications) | 9 | 3
Nonpump thrombus related (Injury, poisoning and procedural complications) | 1 | 0
Minor device malfunction (Injury, poisoning and procedural complications) | 2 | 0
Hemolysis (Blood and lymphatic system disorders) | 4 | 2
Localized nondevice infection (Infections and infestations) | 20 | 14
Sepsis (Infections and infestations) | 14 | 6
Percutaneous site and/or pocket infection (Infections and infestations) | 6 | 5
Toxic metabolic encephalopathy (Nervous system disorders) | 5 | 4
Ischemic stroke (Nervous system disorders) | 6 | 1
Intracranial hemorrhage (Nervous system disorders) | 6 | 0
Transient ischemic attack (Nervous system disorders) | 3 | 1
Other neurological dysfunction (Nervous system disorders) | 5 | 3
Renal dysfunction (Renal and urinary disorders) | 10 | 5
Right heart failure (Cardiac disorders) | 19 | 10
Potential Inflammatory Responses (General disorders) | 1 | 0
Pericardial Fluid Collection (Cardiac disorders) | 8 | 3
Vasodilatory State (Cardiac disorders) | 3 | 0
Hepatic Dysfunction (Hepatobiliary disorders) | 1 | 1
Hypertension (Vascular disorders) | 4 | 1
MI (Non-perioperative) (Cardiac disorders) | 1 | 0
Psychiatric Episode (Psychiatric disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Arterial Non-CNS Thromboembolism (Vascular disorders) | 1 | 0
Venous Thromboembolism Event (Blood and lymphatic system disorders) | 2 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Sustained SVT dysrhytmia (Cardiac disorders) | 14 | 3 — Sustained supraventricular dysrhythmia requiring drug treatment or cardioversion
Localized nondevice infection (Infections and infestations) | 16 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MPC Intramyocardial Injection (N=106) | Control Solution (N=53)
Sustained supraventricular dysrhythmia (Cardiac disorders) | 14 | 3 — Sustained supraventricular dysrhythmia requiring drug treatment or cardioversion
Localized nondevice infection (Infections and infestations) | 16 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02362646/Prot_SAP_000.pdf